CLINICAL TRIAL: NCT02639481
Title: Erigo®Pro Coma Outcome Study - Study on the Effectiveness of a Robotic Tilt Table Device for Recovery of Consciousness
Acronym: EriCOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Therapiezentrum Burgau (Other)
Responsible Party: Principal Investigator, Andreas Bender, Professor of Neurology, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 560-15
Record Dates: First submitted 2015-12-22; First posted 2015-12-24 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Brain Injuries; Disorders of Consciousness
Keywords: traumatic brain injury; stroke; disorders of consciousness; rehabilitation; robotic rehabilitation device
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders; Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group standard physiotherapy (Active Comparator): Patients will receive standard physiotherapy for 60 minutes, including the goal of verticalization and stimulation of the patient but without the use of the robotic Erigo®Pro device.
  Interventions: Behavioral: Standard physiotherapy
- Erigo®Pro group without FES (Active Comparator): Patients will receive 60 minutes of therapy with the robotic Erigo®Pro verticalization device but without functional electrical stimulation (FES) of the leg muscles.
  Interventions: Device: Erigo®Pro group without FES
- Erigo®Pro group with FES (Active Comparator): Patients will receive 60 minutes of therapy with the robotic Erigo®Pro verticalization device including functional electrical stimulation (FES) of the leg muscles.
  Interventions: Device: Erigo®Pro group with FES

INTERVENTIONS:
Behavioral: Standard physiotherapy — Classical standard physiotherapy, including measures to verticalize patients by means of orthesis, classical tilt tables, or castings
  Arms: Control group standard physiotherapy
Device: Erigo®Pro group without FES — Use of the Erigo®Pro device to verticalize patients to above 60° while performing robotic stepping leg movements. FES ist not used.
  Arms: Erigo®Pro group without FES
Device: Erigo®Pro group with FES — Use of the Erigo®Pro device to verticalize patients to above 60° while performing robotic stepping leg movements. FES is applied during then whole treatment session, providing electrical stimulation to the muscles of the upper and lower leg, synchronous to the robotic stepping movements
  Arms: Erigo®Pro group with FES

SUMMARY:
Patients with acquired brain injury (ABI) often suffer from severe disorders of consciousness (DOC), such as coma, unresponsive wakefulness syndrome (UWS), or minimally conscious state (MCS). This study examines the effect, a novel robotic rehabilitation device (the Erigo®Pro system) has on the recovery of consciousness of DOC patients. The device enables patients to be verticalized very early during acute neurorehabilitation and includes robotic leg movement training as well as functional electrical stimulation (FES) of leg nerves. Patients will be randomly allocated to one of three treatment groups: (i) control group with standard physiotherapy without the device, (ii) device treatment without FES, and (iii) device treatment with FES. Time until recovery of consciousness, rehabilitation outcome, and amount of complications will be the outcome variables.

DETAILED DESCRIPTION:
Patients with acquired brain injury (ABI) often suffer from severe disorders of consciousness (DOC), such as coma, unresponsive wakefulness syndrome (UWS), or minimally conscious state (MCS). These DOC can be temporary or persistent. Verticalization and multisensory stimulation are traditionally important therapeutic principles in the neurorehabilitation of such patients. These principles have not yet been tested in randomized controlled trials yet. This trial will therefore evaluate the effect that a 4 week training with a verticalization device (the Erigo®Pro system) with integrated repetitive robotic leg movements and functional electrical stimulation of the leg muscles (FES) has on the clinical course of DOC patients in an inpatient neurorehabilitation setting, following acute ABI. 156 patients will be randomized 1:1:1 to one of the following groups: (i) control group without the Erigo®Pro, (ii) treatment with the Erigo®Pro without FES, and (iii) treatment with the Erigo®Pro and simultaneous FES. There will be 4 training sessions per week for 4 weeks with each session being 60 minutes in length. This will be part of the standard neurorehabilitation program, which in Germany comprises 300 minutes of therapy per day. Patients in the active treatment groups ii) and iii) are required to be verticalized above 60° for at least 35 minutes per treatment session. Patients in the control group will be treated with conventional methods, including verticalization by therapists but without the help of the device. FES will be conducted with the following parameters: 8 channels covering the major ventral and dorsal muscles of the upper and lower, initial current 10 milli ampere (mA), pulse with 250 micro seconds (µs), frequency 25 herz (Hz), ramp 3. Current will be gradually increased to the motor threshold plus 20%.

The investigators will test the following hypotheses:

1. Treatment with the Erigo®Pro system will lead to a quicker recovery of consciousness (increase of at least one diagnostic category of the CRS-R) than conventional therapy,
2. Treatment with the Erigo®Pro system including FES will lead to a quicker recovery of consciousness than using the Erigo®Pro without FES, 3).) Treatment with the Erigo®Pro system will decrease spasticity and complications of neurorehabilitation (pneumonia, pressure ulcers) than conventional therapy, and

4.) Treatment with the Erigo®Pro system will lead to an improved longterm patient outcome (6 months) with regard to independence in the activities of daily living, compared to conventional therapy.

The main outcome variable is the Coma Recovery Scale - revised (CRS-R), secondary variables are the Functional Independence Measure (FIM), the Nociception Coma Scale (NCS), the Modified Ashworth Scale for spasticity, and quantitative HD-EEG measures for brain activity (power, variability, entropy).

Study visits will be prior to first treatment (t0), during the first treatment in vertical position (t1), directly following the first treatment in horizontal patient positioning (t2), 2 weeks after the first treatment (halfway through treatment protocol, t3), at the end of the final treatment after weeks (t4), and final outcome measurement, 6 months after the patient inclusion (t5) within the patients living environment (nursing home or home).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided by legal representative of patient
* unresponsive wakefulness syndrome (UWS) or minimal conscious state (MCS), defined by CRS-R
* acquired brain injury as reason for disorder of consciousness

Exclusion Criteria:

* pre-existing coma, UWS, or MCS
* permanent sedation and/or analgesia with continuous i.v.-application
* body weight > 135 kg
* length of leg of less than 75 cm or more than 100 cm
* contractures in leg joints
* unstable fractures
* open wounds / severe skin irritations on the leg
* severe heart failure or unstable arrhythmias
* aggressive / uncooperative behavior
* other medical reasons for strict bed rest
* severe arterial occlusion disease of the legs
* cardiac pacer
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Time to recovery of consciousness | 4 weeks
  Time to improve 1 diagnostic consciousness category in the Coma Recovery Scale - Revised (CRS-R)

SECONDARY OUTCOMES:
Independence in the activities of daily living | 6 months
  How independent are patients 6 months after study inclusion, measured by the Functional Independence Measure (FIM)
Degree of spasticity | 4 weeks
  Degree of spasticity, measured with the modified Ashworth Scale (mAS)
Occurrence of typical neurorehabilitation complications | 4 weeks
  Do pneumonias and pressure ulcers occur in a patient (clinical observation)?
Change in bioelectrical brain activity | 4 weeks
  Does treatment lead to increased bioelectrical brain activity, measured by high density EEG (power, variability, entropy)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bender, Prof.Dr., Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (2):
- Germany (2):
  - Therapiezentrum Burgau, Burgau, Bavaria
  - Department of Neurology, University of Munich, Munich, Bavaria

REFERENCES:
- [Derived] Rosenfelder MJ, Helmschrott VC, Willacker L, Einhaupl B, Raiser TM, Bender A. Effect of robotic tilt table verticalization on recovery in patients with disorders of consciousness: a randomized controlled trial. J Neurol. 2023 Mar;270(3):1721-1734. doi: 10.1007/s00415-022-11508-x. Epub 2022 Dec 19. PMID 36536249